CLINICAL TRIAL: NCT00901108
Title: Prospective Randomized Controlled Trial of Trabectome Versus Trabeculectomy With Mitomycin C in Patients With Open Angle Glaucoma
Brief Title: Trabectome Versus Trabeculectomy With Mitomycin C in Patients With Open Angle Glaucoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow study recruitment and lack of clinical equipoise over time
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Karim Damji, Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAKD-001
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Open Angle Glaucoma
Keywords: open angle glaucoma; trabectome; trabeculectomy; cataract
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trabectome-IOL (Active Comparator): Combined Trabectome and cataract extraction with intraocular lens insertion
  Interventions: Procedure: Trabectome-IOL
- Trab-IOL (Active Comparator): Combined Trabeculetomy with Mitomycin C and cataract extraction with intraocular lens insertion
  Interventions: Procedure: Trab-IOL

INTERVENTIONS:
Procedure: Trabectome-IOL — Trabectome removes an arc of trabecular meshwork and inner wall of Schlemm's canal to enhance aqueous outflow through natural drainage pathways.
  Trabectome will be done first, followed by cataract surgery because Trabectome requires a clear view through the cornea using a goniolens, and this view may be compromised after cataract surgery.
  Arms: Trabectome-IOL
Procedure: Trab-IOL — Trabeculectomy bypasses the normal aqueous outflow channels of the eye and creates an external filtration pathway (called a filtering bleb) for aqueous to drain and be reabsorbed back into the circulation. Mitomycin C is an agent used during this procedure to decrease scar formation around the new passage.
  Cataract surgery will be done first, followed by Trabeculectomy with Mitomycin C.
  Arms: Trab-IOL

SUMMARY:
The purpose of this study is to compare the efficacy and safety of Trabectome versus Trabeculectomy with adjunctive Mitomycin C, combined with cataract surgery, in patients with open angle glaucoma.

DETAILED DESCRIPTION:
Background: Trabeculectomy with adjunctive use of Mitomycin C (Trab MMC) is the standard incisional procedure to lower intraocular pressure (IOP) in adults with open angle glaucoma (OAG). Trab MMC has been shown to effectively lower IOP, however, it can be associated with a number of serious complications, such as hypotony maculopathy, choroidal effusion or hemorrhage, and endophthalmitis, as well as less serious complications that may affect vision related quality of life such as bleb dysesthesia.

A newer technology, referred to as the Trabectome (NeoMedix Corp., San Juan Capistrano, CA), removes an arc of trabecular meshwork and inner wall of Schlemm's canal with microcautery and appears to lower IOP effectively with fewer and less serious complications than Trab MMC. However, more studies are needed to determine the long term safety and efficacy of this relatively new procedure.

In addition, for OAG patients with visually significant cataracts, either Trab MMC or Trabectome can be combined with cataract surgery.

Study Objective: To compare the efficacy and safety of Trabectome versus Trab MMC, in combination with cataract extraction by phacoemulsification and intraocular lens implant, for control of IOP in OAG, including pseudoexfoliative glaucoma.

Methods: Single center, single surgeon, prospective randomized controlled trial. A total of 52 eligible participants, 26 per study arm would need to be recruited for 90% power. One eye per study patient will be enrolled and randomized to Trabectome combined with cataract surgery (Trabectome-IOL) or Trab MMC combined with cataract surgery (Trab-IOL).

Postoperative visits will take place at the discretion of the surgeon but will include at least visits at day 1, week 1, and months 1, 3, 6, and 12. Postoperative glaucoma medications will be added in a stepped regimen as appropriate, along with additional laser or surgical procedures if needed.

Current Study Status: The clinical trial was terminated early due to slow recruitment and clearer indications for each technique over time leading to lack of clinical equipoise essential for patient randomization/recruitment. This had been discussed and agreed upon with our data safety monitoring board. A total of 19 participants were recruited with followup to one year. Study analysis is pending.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-85 years
2. Open angle glaucoma (including pseudo exfoliative glaucoma)
3. Open angles (≥ Shaffer grade II)
4. Inadequately controlled IOP requiring surgical intervention
5. Visually significant cataract
6. Willing to complete quality of life questionnaires
7. Capable of informed consent and available for at least 1 year follow-up

Exclusion Criteria:

1. Any form of angle closure glaucoma
2. Secondary open angle glaucomas
3. Absence of clear angle landmarks on gonioscopy
4. Other ocular disease that may affect assessments of visual acuity, visual field, or accurate tonometry
5. Previous angle surgery or filtering procedure
6. Steroid use within the preceding 3 months
7. Presence of significant co-morbidities

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-11; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Mean IOP at 6 months | 6 months
Surgical complication rates | intraoperative and postoperative up to 12 months

SECONDARY OUTCOMES:
Mean difference in IOP from baseline to 6 months | 6 months
Mean IOP at 12 months | 12 months
Quality of life measures | preoperative and postoperative at 6 and 12 months
Mean number of glaucoma medications | 12 months
Visual acuity | 12 months
Need for additional laser (excluding suture lysis) and surgical interventions | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karim F Damji, MD FRCSC MBA, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu K, Shah A, Virgili G, Bunce C, Gazzard G. Ab interno trabecular bypass surgery with Trabectome for open-angle glaucoma. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD011693. doi: 10.1002/14651858.CD011693.pub3. PMID 33580495
- [Derived] Hu K, Gazzard G, Bunce C, Wormald R. Ab interno trabecular bypass surgery with Trabectome for open angle glaucoma. Cochrane Database Syst Rev. 2016 Aug 15;(8):CD011693. doi: 10.1002/14651858.CD011693.pub2. PMID 27526051